CLINICAL TRIAL: NCT04109027
Title: Strengthening Neuro-Cognitive Skills for Success in School, Work and Beyond
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N3141-R
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: TBI; Cognitive Dysfunction
Keywords: attention; working memory; executive functioning
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized trial with two active comparison interventions
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Outcomes assessors and investigators will be blinded to study arm. Participants will have equal expectations of learning and benefit from the two active comparisons, though they cannot be blinded to the content of the training interventions. Trainers will have to be aware of the training content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BrainStrong-GSR (Experimental): Goal-directed State Regulation Training (GSR)
  Interventions: Behavioral: BrainStrong-GSR
- BrainStrong-OPT (Active Comparator): Optimization of Brain Functioning (OPT)
  Interventions: Behavioral: BrainStrong-OPT

INTERVENTIONS:
Behavioral: BrainStrong-GSR — Goal-directed State Regulation Training (GSR)
  Other Names: Goal-directed State Regulation Training (GSR)
  Arms: BrainStrong-GSR
Behavioral: BrainStrong-OPT — Optimization of Brain Functioning (OPT)
  Other Names: Optimization of Brain Functioning (OPT)
  Arms: BrainStrong-OPT

SUMMARY:
For many Veterans, success in achieving goals at work, school and in other aspects of life are top priorities. The abilities to regulate attention, remember key information, and stay calm and on track are fundamental to this success. Unfortunately, Veterans who have experienced a traumatic brain injury (TBI) often struggle with these very abilities, and a number of barriers can make it difficult for them to access the help Veterans need. Tele-rehabilitation has the potential to overcome some of these barriers and increase access to care, enabling providers to better reach Veterans 'where they are' in their communities. This project will assess two different approaches to brain injury rehabilitation that seek to help Veterans build personal strengths to better accomplish their goals. Both approaches will be delivered remotely via tele-rehabilitation and augmented by digital apps to best support Veterans' learning in community settings outside the VA.

DETAILED DESCRIPTION:
This project will offer two training approaches targeting difficulties with goal-directed functioning associated with traumatic brain injury. Both approaches will be delivered remotely via tele-rehabilitation and augmented by digital apps - an intervention framework that addresses known barriers to engagement (e.g., convenience and access) and provides tools to intensify training. The study will be open to eligible Veterans (ages 21-60 years old) with history of mild-to-moderate TBI who experience difficulties with cognitive-emotional regulation and goal-directed functioning. After screening for eligibility and providing informed consent, participants will be allocated by permuted block randomization into one of two treatments: Education to optimize brain functioning (OPT), which will teach Veterans about brain health, brain injury and factors that affect brain functioning, or training in goal-directed state regulation skills (GSR), which will teach Veterans skills for regulating cognitive-emotional functioning during goal pursuit. A special emphasis on outreach will be to recruit student Veterans with TBI.

Each intervention will be matched for delivery method, expectation of benefit, workload and attention, and overall duration. Training will last approximately five weeks, accommodating typical academic schedules. Participants will undergo multi-level assessments at baseline (prior to interventions), immediately after training, and at 3 months follow-up, administered in-person by staff at study sites. In order to investigate effects on goal-directed functioning at multiple levels, assessments will include (1) measures of performance on neurocognitive tasks; (2) functional performance on complex, goal-based tasks; (3) ratings of changes in functioning in personal life, and (4) progress toward personal goals as measured with goal attainment scaling procedures. Data will be analyzed to assess immediate and long term changes associated with each intervention; immediate and long-term differences between the interventions; and moderators and mediators of intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Post 9/11 Veterans
* age 21-60; with history of mild-moderate TBI (including reported mechanism of head injury and alteration of consciousness);
* in the chronic, stable phase of recovery (>6 months from injury); with at least 1 self-reported cognitive symptom, --including difficulties with working memory; and interested in goal-setting and intensive training.

Exclusion Criteria:

* Severely apathetic/abulic, aphasic, or other reasons for being unable or unwilling to participate in training;
* severe cognitive dysfunction (below 2 standard deviations on two composite cognitive domains);
* schizophrenia;
* bipolar disorder;
* history of other neurological disorders;
* current medical illnesses that may alter mental status or disrupt participation in the study;
* active psychotropic medication changes;
* symptom magnification or malingering.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Selective Information Processing | Change from baseline to 2 weeks post-intervention
  In order to test a primary hypothesis related to potential intervention mechanisms, the investigators will use the well-established Automated Operation Span Task (OSPAN) to measure working memory in the presence of distractions. Specifically, the OSPAN sums correctly recalled and ordered items from a memory set in the presence of distractors. The investigators elected to use this psychometric measure due to its sensitivity, precision, and test-retest stability in order to maximize the ability to detect longitudinal changes on the primary outcome of interest.

SECONDARY OUTCOMES:
Observed Functional performance | 2 weeks post-intervention, 3 months post-intervention
  The Goal Processing Scale (GPS) measures goal-directed functioning in a complex, ecologically-valid setting. This timed procedure requires participants gather information on three different self-selected activities. Throughout the task, participants are required to follow specific rules and manage unanticipated challenges (e.g., distractions). Evaluators, following a well-specified manual, rate participants' performance across multiple domains of functioning (e.g., maintaining attention in a distracting environment, cognitive flexibility) while they complete the task. The outcome variable of interest will be changes to the GPS total score. GPS scores range from 0 - 10, with higher scores reflecting better goal-directed functioning. Positive change scores will reflect pre-post training improvements to goal-directed functioning, with negative change scores reflecting pre-post worsening of goal-directed functioning.
Progress Towards Goal Attainment | 3 months post-intervention
  Goal Attainment Scaling (GAS) procedures will be used for setting and measuring progress toward participant goals. GAS is a six-step process to quantify clinically meaningful change. GAS is a highly individualized but quantitative outcome measure. Participants will define goals to complete and identify objective and observable outcomes for each goal, consisting of outcomes both better and worse than anticipated. Participants weigh goals based upon their estimated difficulty level and priority. GAS scores range from -2 to +2, with negative scores indicating participants achieved less than expected, a score of "0" indicating that participants achieved at expectation, and positive scores indicating that participants scored better than expected. The outcome of interest will be the weighted average of each GAS score evaluated post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J. W. Chen, MD MA, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No